CLINICAL TRIAL: NCT01974492
Title: A Comparison of Histologic and Immunohistochemical Characteristics Between the Upper and Lower Leg Saphenous Veins Used for Coronary Artery Bypass Grafting
Brief Title: Comparison of Saphenous Vein Graft Harvested From Upper Versus Lower Leg in Coronary Artery Bypass Grafting
Acronym: COSAVEGUL-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ki-Bong Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUHTS_KBKim_Saphenous
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Triple Vessel Disease; Unstable Angina; Stable Angina; Myocardial Infarction
Keywords: saphenous vein graft; composite graft; coronary artery bypass grafting; graft remodeling
MeSH Terms: conditions — Angina, Unstable; Angina, Stable; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Upper leg vein (Active Comparator): Upper leg vein harvesting
  Interventions: Procedure: Upper leg vein harvesting
- Lower leg vein (Active Comparator): Lower leg vein harvesting
  Interventions: Procedure: Lower leg vein harvesting

INTERVENTIONS:
Procedure: Upper leg vein harvesting — Patients whose saphenous veins are harvested from upper legs.
  Arms: Upper leg vein
Procedure: Lower leg vein harvesting — Patients whose saphenous veins are harvested from lower legs.
  Arms: Lower leg vein

SUMMARY:
In coronary artery bypass grafting, saphenous veins are widely used as a composite grafts that are Y-anastomosed to in-situ left internal thoracic artery. Based on our observation that remodeling of saphenous vein graft differs between those harvested from upper leg vein and lower leg, this study aims to compare histologic and immunohistochemical findings between saphenous vein grafts harvested from upper leg and lower leg.

DETAILED DESCRIPTION:
Inclusion criteria:

* Patients aged from 40 to 75 years with triple vessel disease
* Patients who are eligible for the use of left internal thoracic artery as an in situ primary conduit
* Operation plan: saphenous vein graft will be Y-anastomosed to left internal thoracic artery.
* Patients whose saphenous vein grafts can be harvested from both upper legs and lower legs
* Patients who are eligible for off-pump coronary artery bypass grafting
* Patients who agreed with the participation in the research based on thorough explanation.

Patients will be randomly assigned to upper leg vein (ULV) group and lower leg vein (LLV) group immediately after anesthetic induction.

Pieces of residual saphenous vein graft will be sent for histologic and immunohistochemical examination for the evaluation of endothelial cell preservation and the expression of matrix proteins.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multivessel disease who were planned to undergo off-pump coronary artery bypass grafting
* Patients whose left internal thoracic arteries can be used, and whose saphenous vein grafts will be Y-anastomosed to left internal thoracic arteries.
* Patients whose saphenous vein grafts can be harvested from both upper and lower legs.

Exclusion Criteria:

* Patients with overt heart failure symptoms
* Patients with intractable ventricular arrhythmia
* Patients with history of cancer or malignancy
* Patients with coagulation or other hematologic disorder
* Patients who needs concomitant cardiac procedures

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Endothelial preservation of saphenous vein graft | 1 year
  Participants will be followed for the duration of hospital stay, an expected average of 1 week.

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Bong Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea